CLINICAL TRIAL: NCT05987254
Title: Comparison Between Peri-Capsular Nerve Group and Supra Inguinal Fascia Iliaca BLOCK for Analgesia and Ease of Positioning During Neuraxial Anesthesia in Hip Fracture Patients: A Randomized Clinical Trial.
Brief Title: Peri-Capsular Nerve Group and Supra Inguinal Fascia Iliaca BLOCK for Analgesia and Ease of Positioning During Neuraxial Anesthesia in Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC 11-3-2023
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Spinal Anesthesia; Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FICB group (Active Comparator): received ultrasound guided suprainguinal fascia iliaca block
  Interventions: Procedure: suprainguinal fascia iliaca block
- PENG group (Active Comparator): received ultrasound guided pericapsular nerve group block
  Interventions: Procedure: pericapsular nerve group block

INTERVENTIONS:
Procedure: suprainguinal fascia iliaca block — ultrasound guided suprainguinal fascia iliaca block
  Arms: FICB group
Procedure: pericapsular nerve group block — ultrasound guided pericapsular nerve group block
  Arms: PENG group

SUMMARY:
Severe pain associated with fractured hip often results in difficulty during positioning for spinal anesthesia (SA). Among many regional analgesic techniques, the fascia iliaca compartment block (FICB) is popular among anesthesiologists to provide immediate as well as postoperative analgesia in hip fractures. Recently, the pericapsular nerve group (PENG) block has been proposed to provide effective analgesia in hip fracture patients. However, comparative studies between PENG and FICB are lacking.

ELIGIBILITY:
Inclusion Criteria:

* 40 years and above with hip fracture with persistent pain and scheduled for surgery under spinal anesthesia (SA)

Exclusion Criteria:

* any contraindications to SA or peripheral nerve blocks, history of ischaemic heart disease, patients on opioids for chronic pain and patients with significant cognitive impairment. Patients who had no pain while sitting by themselves (resting pain less than 4 on NRS) for SA without any support were also excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
NRS | 30 minute postoperative
  In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
The ease of spinal positioning (EOSP) | Thirty minutes after the blocks
  The ease of spinal positioning (EOSP) was assessed on the scale of 0-3 (0 = unable to position, 1 = patient had abnormal posturing due to pain and required support for positioning, 2 = mild discomfort but does not require support for positioning, 3 = optimal condition where the patient was able to position himself without pain)

SECONDARY OUTCOMES:
amount of tramadol used | 24 hours postoperatively
  number of rescue doses of tramadol will be recorded

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Haney Baumey, Banhā
  - Facualty of Pharmacy, Al Azhar University, Cairo
  - Neveen Kohaf, Tanta

IPD SHARING:
Plan to Share IPD: Yes
data will be shared upon resealable request from the principal investigator
Supporting Information: Study Protocol, SAP